CLINICAL TRIAL: NCT03084861
Title: A Multicenter, Randomized, Open-label, Two-arms Phase I/II Clinical Trial to Asses Efficacy and Safety of Cord Blood Eye Drops in Neurotrophic Keratopathy
Brief Title: A Clinical Trial to Asses Efficacy and Safety of Cord Blood Eye Drops in Neurotrophic Keratopathy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low recruitment. No safety issue associated.
Sponsor: Banc de Sang i Teixits (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I.2016.010
Record Dates: First submitted 2017-03-08; First posted 2017-03-21 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Neurotrophic Keratopathy

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cord blood eye drops (Experimental): Experimental drug: cord blood eye drops Description: eye drops plasma from cord blood diluted v/v with Plasmalyte®, without antimicrobial preservatives Dosage regimen: 1 drop every 2 hours Pharmaceutical form: ophthalmic preparation eye drops Presentation: batch of 19 vials of 1 mL per vial Route of administration: ophthalmic/ocular
  Interventions: Drug: Cord Blood Eye Drops
- Conventional treatment (Active Comparator): Conventional treatment:
  1. Artificial tears Description: Lubristil ® (single dose) Dosage regimen: 1 drop every 2 hours Pharmaceutical form: ophthalmic preparation eye drops Presentation: batch of 20 or 30 vials of 0.3 mL per vial Route of administration: ophthalmic
  2. Therapeutic Contact lens Description: Air Optix Night&Day Dosage regimen: 1 contact lens per visit Pharmaceutical form: contact lens Presentation: 1 unit per case Route of administration: ophthalmic/ocular
  Interventions: Drug: Conventional treatment

INTERVENTIONS:
Drug: Cord Blood Eye Drops — Eye drops plasma from cord blood diluted v/v with Plasmalyte®, without antimicrobial preservatives
  Arms: cord blood eye drops
Drug: Conventional treatment — 1. Artificial tears: Lubristil ®
  2. Therapeutic Contact lens: Air Optix Night&Day
  Arms: Conventional treatment

SUMMARY:
This is a multicenter, randomized, open-label, two-arms phase I/II, clinical trial, in which 42 patients will be enrolled with the principal objective to evaluate the efficacy through changes in lesion size and, secondary, to evaluate the safety and efficacy through corneal sensibility, corneal opacity, visual acuity and complications of Neurotrophic Keratopathy (NK). Patients will be randomized 1:1 to receive experimental treatment (cord blood eye drops) or conventional treatment (artificial tears and therapeutic contact lens).

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, two-arms phase I/II, clinical trial, in which 42 patients will be enrolled with the principal objective to evaluate the efficacy through changes in lesion size and, secondary, to evaluate the safety and efficacy through corneal sensibility, corneal opacity, visual acuity and complications of NK. Patients will be randomized 1:1 to receive experimental treatment (cord blood eye drops) or conventional treatment (artificial tears and therapeutic contact lens).

All patients, with conventional or experimental treatment, will be treated for 19 days. A topical antibiotic will be added too as a concomitant treatment to all treatment groups, until the injury closes or according to medical criteria.

After signing informed consent, inclusion and exclusion criteria will be assessed, and if the patient meets all the requirements, the patient will be randomized.

After initiation of the treatment, patients will be follow-up at 2-3 days and once a week for 3 weeks. A final follow-up is planned at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. NK stage 2 or 3 (Mackie classification)
3. Signed Informed Consent Form
4. The patient is able to understand the nature of the study and to participate throughout its duration

Exclusion Criteria:

1. Medical history of eye tumors
2. Active eye infection
3. Eyelid bad position or eyelid closure problems
4. Conjunctiva scarring
5. Topic chronic eye treatments with corticoids
6. Acute corneal burns (<3 months)
7. Intolerance to contact lens
8. Allergy or inability to receive concomitant treatment with Exocin®
9. Patients with immunosuppressive or chemotherapy treatment
10. Pregnant woman or woman without proper contraceptive methods according to the investigator (*), or lactating women
11. Participation in another clinical trial in the last month (*) Contraceptive methods accepted in the protocol are: hormonal, intrauterine device (IUD), barrier methods, voluntary sterilization or the patient has menopause >1 year duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Corneal lesion size | after 3 weeks post-treatment,
  Variation percentage in corneal lesion size

SECONDARY OUTCOMES:
Incidence of Adverse Events | From date of randomization until the date of the last visit (6 weeks post-treatment)
  Safety evaluation through laboratory data and adverse events
Corneal lesion size | at 2-3 days post-treatment and at 1, 2 and 6 weeks post-treatment
  Variation percentage in corneal lesion size
Stage on the corneal lesion | at 3 weeks post-treatment
  Changes stage on the corneal lesion (cured, stage 1, stage 2, stage 3) from baseline
Qualitative scale of corneal sensibility | at 2-3 days post-treatment and at 1, 2, 3 and 6 weeks post-treatment
  Changes in qualitative scale of corneal sensibility (normoesthesia, hypoesthesia, anesthesia)
Corneal opacity | at 2-3 days post-treatment and at 1, 2, 3 and 6 weeks post-treatment
  Changes on corneal opacity from baseline (not response, improvement, worse)
Visual acuity | at 2-3 days post-treatment and at 1, 2 and 6 weeks post-treatment
  Line variation in relation to visual acuity
Neurotrophic keratopathy | From date of randomization until the date of the last visit (6 weeks post-treatment)
  Number of neurotrophic keratopathy complications

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Querol Giner, MD PHD, Principal Investigator — Banc de Sang i Teixits
Locations (10):
- Spain (10):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Mútua de Terrassa, Terrassa, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Instituto Oftalmológico Quirónsalud Barcelona, Barcelona
  - Hospital de l'Esperança, Barcelona
  - Institut de microcirurgia ocular IMO, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Josep Trueta, Girona
  - Hospital Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samarkanova D, Martin S, Bisbe L, Puig J, Calatayud-Pinuaga M, Rodriguez L, Azqueta C, Coll R, Casaroli-Marano R, Madrigal A, Rebulla P, Querol S; Barcelona CBED Study Group (Appendix I). Clinical evaluation of allogeneic eye drops from cord blood platelet lysate. Blood Transfus. 2021 Jul;19(4):347-356. doi: 10.2450/2020.0130-20. Epub 2020 Oct 9. PMID 33085593